CLINICAL TRIAL: NCT02476058
Title: An Exploratory Multicenter, Double-Blind, Diphenhydramine- and Placebo-Controlled Safety, Efficacy and Biomarker Study With JNJ-42847922 in Subjects With Major Depressive Disorder
Brief Title: A Safety, Efficacy and Biomarker Study of JNJ-42847922 in Participants With Major Depressive Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR107002; 42847922MDD1001 (Other: Janssen-Cilag International NV); 2014-005182-75 (EudraCT Number)
Record Dates: First submitted 2015-05-29; First posted 2015-06-19 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; JNJ-42847922; Diphenhydramine; Placebo
MeSH Terms: conditions — Depressive Disorder, Major | interventions — seltorexant; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (3):
- JNJ-42847922 (Experimental): JNJ-428479, 20 milligram (mg) capsule, orally, once daily, at bedtime for 10 days in women of childbearing potential (WOCBP) or for 4 weeks in all other participants.
  Interventions: Drug: JNJ-42847922
- Diphenhydramine (Experimental): Diphenhydramine 25 mg capsule, orally, once daily, at bedtime for 10 days in women of childbearing potential (WOCBP) or for 4 weeks in all other participants.
  Interventions: Drug: Diphenhydramine
- Placebo (Placebo Comparator): Matching placebo (capsules containing neutral pellets), orally, once daily, at bedtime for 10 days in women of childbearing potential (WOCBP) or for 4 weeks in all other participants.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-42847922 — JNJ-428479, 20 milligram (mg) capsule, orally, once daily, at bedtime for 10 days in women of childbearing potential (WOCBP) or for 4 weeks in all other participants.
  Arms: JNJ-42847922
Drug: Diphenhydramine — Diphenhydramine 25 mg capsule, orally, once daily, at bedtime for 10 days in women of childbearing potential (WOCBP) or for 4 weeks in all other participants.
  Arms: Diphenhydramine
Drug: Placebo — Matching placebo (capsules containing neutral pellets), orally, once daily, at bedtime for 10 days in women of childbearing potential (WOCBP) or for 4 weeks in all other participants.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of JNJ-42847922 in participants with Major Depressive Disorder (MDD).

DETAILED DESCRIPTION:
This will be a multi-center (when more than one hospital works on a medical research study), randomized (study medication assigned to participants by chance), double-blind (neither the researchers nor the participants know what treatment the participant is receiving) and placebo-controlled (an inactive substance; a pretend treatment [with no drug in it] that is compared in a clinical trial with a drug to test if the drug has a real effect) study. This study will consist of an eligibility screening examination (between 28 days and 1 day prior to the first dose administration), a parallel group treatment phase of 10 days or 4 weeks, and a follow-up period of 2 weeks including 2 follow-up visits. The duration of study will be 12 months. Participants will be randomly assigned to receive either JNJ-42847922, Diphenhydramine or Placebo. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Before randomization, a woman must be either: 1) Not of childbearing potential: postmenopausal; permanently sterilized; or otherwise be incapable of pregnancy. 2) Of childbearing potential and practicing a highly effective method of birth control consistent with local regulations regarding the use of birth control methods for participants participating in clinical studies: example, established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device (IUD) or intrauterine system (IUS) in combination with barrier methods: condom with spermicidal foam/gel/film/cream/suppository or occlusive cap with spermicidal foam/gel/film/cream/suppository; male partner sterilization; true abstinence. Women must agree to continue using these methods of contraception throughout the study and for at least 3 months after receiving the last dose of study medication
* Participant Body mass index (BMI) must be between 18 and 30 kilogram per square meter (kg/m2) inclusive
* Participant must meet the Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) or 5 diagnostic criteria for major depressive disorder (MDD) without psychotic features, and confirmed by the Mini International Neuropsychiatric Interview (MINI) 6.0; Participant must have an Inventory of Depressive Symptomatology- Clinician rated-30 (IDS-C30) total score greater than or equal to (>=) 30; Participant is either currently antidepressant naive or currently being treated with a maximum of two concurrent antidepressants. If the subject is currently treated with antidepressants, they have to be given at an optimal dose and for at least 4 weeks, but not longer than 24 weeks with a suboptimal response
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control e.g., either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Participant must be willing and able to adhere to the prohibitions and restrictions specified in this protocol

Exclusion Criteria:

* Women who is pregnant or breast feeding
* Participant has a history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the investigator, with concurrence with the sponsor's study responsible physician, is considered cured with minimal risk of recurrence)
* Participant has a primary DSM diagnosis of general anxiety disorder (GAD), panic disorder, obsessive compulsive disorder (OCD), posttraumatic stress disorder (PTSD), anorexia nervosa, or bulimia nervosa. Subjects with comorbid GAD, social anxiety disorder (SAD), or panic disorder for whom MDD is considered the primary diagnosis are not excluded
* Participant has a length of current major depressive episode (MDE) >24 months despite adequate treatment
* Participant has failed more than 2 treatments with a different pharmacological mode of action despite an adequate dose and duration during a previous, or the current depressive episode

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-06-11 (Actual); Primary Completion 2016-01-04 (Actual); Study Completion 2016-01-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs) | Screening until follow-up phase (up to 12 months)
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; lifethreatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

SECONDARY OUTCOMES:
Participants Leeds Sleep Evaluation Questionnaire (LSEQ) Score | Day 2, 11, 29, 31, 42
  The LSEQ comprises 10 self-rating 100 millimeter (mm)-line analogue questions regarding changes in the quality of sleep and early morning behavior, following any given intervention. Scores range between 0 and 100. Scores beneath 50 indicate better sleep.
Computerized Cognitive Test Battery: ISLT (Verbal Learning and Memory) Test | Day 1, 2 , 5, 6, 10 and 11
  The ISLT is a measure of verbal learning and memory and uses a well-validated list-learning paradigm. The task is administered using a computer. High frequencies, high imagery, concrete nouns (items from a shopping list) are read to the participant by the test supervisor at the rate of one word every two seconds. Once the [12] words have been read, the participant is asked to recall as many of the words as he/she can as quickly as possible. The test supervisor uses a mouse or stylus to mark the words recalled by the participant on the computer screen. When the participant can recall no more words, the same list is read a second time. The test supervisor records the words recalled by the participant on this trial. This is then repeated a third time. The delayed recall condition requires the participant to recall the words from the list after a delay without having the list read again.
Computerized Cognitive Test Battery: Detection (DET) Test | Day 1, 2 , 5, 6, 10 and 11
  Simple reaction time task measuring processing speed; mean of the log10 transformed reaction times for correct responses (lower score = better performance).
Computerized Cognitive Test Battery: Identification (IDN) Test | Day 1, 2 , 5, 6, 10 and 11
  Choice reaction time paradigm measuring attention; mean of the log10 transformed reaction times for correct responses (lower score = better performance).
Computerized Cognitive Test Battery: One Back (OBK) Test | Day 1, 2 , 5, 6, 10 and 11
  Working memory measure; mean of the log10 transformed reaction times for correct responses (lower score = better performance).
Computerized Cognitive Test Battery: Groton Maze Learning Test (GMLT) | Day 1, 2 , 5, 6, 10 and 11
  Executive function measure; total number of errors made in attempting to learn the same hidden pathway on five consecutive trials during a single session (lower score = better performance).
Polysomnography (PSG) Objective Assessment of Latency To Persistent Sleep | Day 1 to 2, 5 to 6 and 10 to 11
  Objective assessment: A central scoring facility was used to derive the PSG sleep parameters Latency to Persistent Sleep (LPS) from the epochs and stages collected via the polysomnography (PSG) recordings. Each epoch is 30 seconds. Latency to persistent sleep (LPS; minutes): time from lights out to the first of 20 consecutive epochs (10 minutes) of non-wake, as determined by PSG recordings.
Subjective Assessment of Latency To Persistent Sleep | Women of childbearing potential (WOCBP): Day 2, 11 and follow up visit (Day 13 and 24); Males and women of non-childbearing potential (WONCBP): Day 2, 11, 29 and follow up visit (Day 31 and 42)
  Subjective assessment: The amount of time measured in minutes it takes to fall asleep was based on participant-reported subjective assessments of sleep disturbance and was obtained from participants' responses to morning questionnaires.
PSG Objective Assessment of Total Sleep Time | Day 1 to 2, 5 to 6 and 10 to 11
  Objective assessment: A central scoring facility was used to derive the PSG sleep parameter of Total Sleep Time (TST) from the epochs and stages collected via the PSG recordings. The PSG parameters provided an objective assessment of the subject's sleep on a given night. Total sleep time was defined as the number of non-wake epochs from the beginning of recording to the end of recording divided by 2.
Subjective Assessment of Total Sleep Time | Women of childbearing potential (WOCBP): Day 2, 11 and follow up visit (Day 13 and 24); Males and women of non-childbearing potential (WONCBP): Day 2, 11, 29 and follow up visit (Day 31 and 42)
  Subjective assessment: The subjective measure was based on participant-reported subjective assessments of sleep disturbance and were obtained from participants' responses to morning questionnaires.
PSG Objective Assessment of Wake Time After Sleep Onset (WASO) | Day 1 to 2, 5 to 6 and 10 to 11
  Objective assessment: A central scoring facility was used to derive the PSG sleep parameters Wake Time After Sleep Onset (WASO) from the epochs and stages collected via the PSG recordings. Each epoch is 30 seconds. Wake time after sleep onset (WASO; minutes): The number of wake epochs after the onset of persistent sleep to the end of the recording, divided by 2.
Subjective Assessment of Wake Time After Sleep Onset (WASO) | Women of childbearing potential (WOCBP): Day 2, 11 and follow up visit (Day 13 and 24); Males and women of non-childbearing potential (WONCBP): Day 2, 11, 29 and follow up visit (Day 31 and 42)
  Subjective assessment: The subjective measure was based on participant-reported subjective assessments and were obtained from participants' responses to morning questionnaires.
Inventory of Depressive Symptomatology-clinician Rated 30 (IDSC30) Score and Structured Interview Guide for Hamilton Depression Scale (SIGH-D) (as combined SIGHD-IDS) | Day 1, 11, 29, 31 and 42
  The SIGHD-IDS is a combined structured interview guide to complete both the structured interview guide for the Hamilton Depression Scale (SIGH-D) and the Inventory of depressive symptomatology (IDS-C30). The SIGH-D interview guide is based on the Hamilton Depression Rating Scale (HDRS17; Williams 1988). It contains 17 items pertaining to symptoms of depression experienced over the past week. Score range is from 0 to 52. The IDS-C30 is a standardized 30 item, clinician rated, scale to assess the severity of a participant's depressive symptoms. The scale uses the 9 symptom domains of the Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV criteria to measure symptom severity. The scores range from a minimum of 0 to a maximum score of 84. The higher the score the more severe the symptoms of depression.
Quick Inventory of Depressive Symptoms-16 (QIDS-SR16) Score | Day 1, 11, 29, 31 and 42
  The QIDS-SR16 is a participant reported measure designed to assess the severity of depressive symptoms. Participants provide responses to each item of this instrument with a 4-point Likert scale, with scores ranging from 0-3 for each item. The 7-day period prior to assessment is the usual recall period for assessing symptom severity. The total score ranges from 0 to 27. Using a scale of severity of depression of none, mild, moderate, severe, and very severe, corresponding QIDS-SR16 total scores are none 1-5, mild 6-10, moderate 11-15, severe 16-20 and very severe 21-27.
Ruminative Response Scale (RRS) Score | Day 1, 11 and 29
  Ruminative Response Scale is used to assess symptoms of rumination. It is a 22-item scale. Each item ranges from 1= almost never to 4 = almost always. Total score ranges from 1 to 4.
Changes in Major Depressive Disorder (MDD)-related Biomarkers | Day 1, 11 and 29
  Different biomarkers in blood (Interleukin-6 [IL-6]) and saliva (cortisol) will be measured to explore a relation to the seriousness of depressive symptoms or exposure to JNJ-42847922.
Plasma concentrations for JNJ-42847922 | Day 1, 2, 6, 11 and 29

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (7):
- Belgium (3):
  - Aalst
  - Brussels
  - Duffel
- Germany (3):
  - Berlin
  - Hamburg
  - Schwerin
- Leiden, Netherlands